CLINICAL TRIAL: NCT02741414
Title: Construction and Application of the Treatment of Refractory Helicobacter Pylori Infection Based on the High-throughput Sequencing Technologies
Brief Title: A Multi-center Study for Eradication of Refractory Helicobacter Pylori
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taizhou Hospital (Other)
Collaborators: Centers for Disease Control and Prevention, China (Other Government); Academy Military Medical Science, China (Industry); First Affiliated Hospital of Zhejiang University (Other); Taizhou Enze Medical Center Group (Other); Taizhou First People's Hospital (Other); The first people Hospital of Linhai (Unknown); Affiliated Wenling Hospital of Wenzhou Medical University (Other); Sanmen People Hospital (Unknown); Xianju People Hospital (Unknown); Tiantai People Hospital (Unknown); Yuhuan People Hospital (Unknown); The second people Hospital of Yuhuan (Unknown); Zhiyuan Medical Inspection Institute (Other)
Responsible Party: Principal Investigator, Liping Ye, Director of the Department of Gastroenterology, Taizhou Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TaizhouH
Record Dates: First submitted 2016-03-25; First posted 2016-04-18 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-03

CONDITIONS: Gastritis
Keywords: Helicobacter pylori; Antibiotic resistance; Sequencing; Mechanism
MeSH Terms: conditions — Gastritis

ARMS (3):
- H pylori culture negative group (Experimental): The patients who have the negative result of H pylori culture were classified into H pylori culture negative group.
  Interventions: Device: The result of H pylori culture based on gram staining and enzyme activity testing
- The first successful eradication group (Experimental): The patients with first eradication therapy of H. pylori infection have the first successful treatment based on the standardized treatment including antibiotics selection from antibiotic susceptibility testing and proton pump inhibitors （PPIs) dose selection from CYP2C19 gene sequencing.
  Interventions: Device: The result of H pylori culture based on gram staining and enzyme activity testing; Device: The result of 13C-urea breath test after treatment based on the selection of clarithromycin, levofloxacin, metronidazole, amoxicillin，tetracycline，furazolidone and the dose of esomeprazole; Device: The result of Amoxicillin resistance in vitro based on antibiotic susceptibility testing
- The refractory infection of H. pylori group (Experimental): The patients with first eradication therapy of H. pylori infection have the two failure treatment based on the standardized treatment including antibiotics selection from antibiotic susceptibility testing and PPIs dose selection from CYP2C19 gene sequencing.
  Interventions: Device: The result of H pylori culture based on gram staining and enzyme activity testing; Device: The result of 13C-urea breath test after treatment based on the selection of clarithromycin, levofloxacin, metronidazole, amoxicillin，tetracycline，furazolidone and the dose of esomeprazole; Device: The result of Amoxicillin resistance in vitro based on antibiotic susceptibility testing

INTERVENTIONS:
Device: The result of H pylori culture based on gram staining and enzyme activity testing — This intervention aimed at patients with the positive result of 13C-urea breath test. Patients with negative result of H pylori culture was H pylori culture negative group. Patients with positive result of H pylori culture were belonged into the first successful eradication group and the refractory infection of H. pylori group.
Device: The result of 13C-urea breath test after treatment based on the selection of clarithromycin, levofloxacin, metronidazole, amoxicillin，tetracycline，furazolidone and the dose of esomeprazole — The intervention focused on the results from the result of 13C-urea breath test after treatment. The first successful eradication group and the refractory infection of H. pylori group were treated according to the antibiotic susceptibility testing and CYP2C19 gene polymorphism. Eight weeks after treatment, a 13C-urea breath test was performed on patients. The first successful eradication group were patients with negative in 13C-urea breath tests in the first treatment. The refractory infection of H. pylori group were treatment failure patients with positive in 13C-urea breath tests after the second standardized treatment.
  Arms: The first successful eradication group; The refractory infection of H. pylori group
Device: The result of Amoxicillin resistance in vitro based on antibiotic susceptibility testing — The intervention focused on the results from the result of Amoxicillin susceptibility testing in vitro. In this study, the investigators selected the patients with Amoxicillin resistance from the first successful eradication group and the refractory infection of H. pylori group.
  Arms: The first successful eradication group; The refractory infection of H. pylori group

SUMMARY:
Recently studies showed that the eradication rate of H. pylori fail to exceed 80% and even falls into an unacceptable range. A major cause of treatment failure is associated with antibiotic resistance and poor patient compliance. However, the refractory infection of H. pylori is still existing, although patients have good compliance and receive standardized treatment. This phenomenon is likely attributed to the different ratio of sensitive and resistance in H. pylori, the difference of Amoxicillin resistance between in vivo and in vitro, the difference between phenotype and genotype or the influence of micro-environment in the stomach. In order to solve the refractory infection of H. pylori, investigators performed a muti-center study together with other 14 institutions. In this study, investigators will select the patients with refractory infection of H. pylori after two standardized treatment from patients with first eradication therapy of H. pylori infection. Then, investigators will perform a high-throughput sequencing for patients in groups. Finally, investigators will compare the differences between the patients with first successful eradication and patients with refractory infection of H. pylori, such as drug resistance gene mutation, phenotype and genotype, the mechanisms of Amoxicillin resistance and micro-environment in stomach.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18~70 years old, male or female, the first eradication therapy of H. pylori infection patients.
2. Symptoms of abdominal pain, bloating, acid efflux, belching, nausea, vomiting, heartburn, chest pain, vomiting, melena, etc.
3. Unused antibiotics, bismuth, H2 receptor antagonists or PPIs by nearly 4 weeks
4. 13C-labelled urea breath test positive.
5. Agreed to Helicobacter pylori culture and sensitivity testing taken by endoscopy gastric biopsy specimens,and the result of culture was positive.
6. Agreed to Helicobacter pylori eradication therapy and cooperate with the eradication efficacy follow-up survey.

Exclusion Criteria:

1. Severe heart, liver, kidney dysfunction.
2. Pregnant or lactating women.
3. Complications of bleeding, perforation, pyloric obstruction, cancer.
4. Esophageal,gastrointestinal surgery history.
5. Patients can not properly express their complaints,such as psychosis, severe neurosis.
6. Taking nonsteroidal antiinflammatory drugs (NSAIDs) or alcohol abusers.
7. Allergic to penicillin or either drugs of the 6 antibiotic tested by susceptibility testing.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4428 (Estimated)
Dates: Start 2016-06; Primary Completion 2018-04 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
The eradication rate of H. pylori reach to 95% in all groups | 1 year
The microflora structure of a total of 240 patients in the first successful eradication group and the refractory infection of H. pylori group | Three months
The proportion of mix infection of H pylori in a total of 240 patients in two groups | Three months
The number of single nucleotide varation（SNV）of 20 patients in the first successful eradication group and the refractory infection of H. pylori group that are related to Amoxicillin resistance | Three months

CONTACTS AND LOCATIONS:
Locations (1):
- Xianju People Hospital, Taizhou, Zhejiang, China